CLINICAL TRIAL: NCT03901443
Title: Survey on Itch in Outpatients of a University Clinic
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: UBE 15/114, sp15Mueller3
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Itch
Keywords: itchy skin diseases; itch treatments; pruriception
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey on itch — self-administered patient questionnaire regarding the different aspects of itch

SUMMARY:
This study is to investigate the pruriception (i.e. the perception of the character and intensity of itch), the impact of itch on quality of life, the response to itch and the subjective efficacy and preferences of the different treatment options among patients with different skin diseases. Better insights into these aspects might help to optimize itch treatment in clinical Settings.

ELIGIBILITY:
Inclusion Criteria:

* outpatients suffering from itch

Exclusion Criteria:

* outpatients (suffering from itch) not willing or able to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All outpatients of the dermatologic university clinic suffering from itch are eligible to participate in the study (from December 2015 until the end of April 2016).
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
itch intensity | single time point assessment at baseline
  Questions regarding itch perception (NRS 0-10; 0 = no itch, 10 = worst imaginable itch) experienced at the moment, within the last 7 days, within the last month
itch perception | single time point assessment at baseline
  Questions regarding situations in which the itch is especially bad (multiple choice options regarding day time, daily situations, season); objective assessment in which respondents are asked to select answers from the choices offered as a list
impact of itch on quality of life | single time point assessment at baseline
  Questions regarding strength of impact of itch on quality of life (NRS 0-10; 0 = no impact, 10 = extreme)
quality of sleep | single time point assessment at baseline
  Questions regarding sleep disturbance by itch (Does itch disturb the patient's sleep and/or sleep of other persons? (yes/no))
days missing at work | single time point assessment at baseline
  Approximate number of days missing at work due to itch within last 6 months
helpfulness of common itch therapies | single time point assessment at baseline
  Questions regarding helpfulness of common itch therapies (NRS 0-10; 0 = no reduction in itch, 10
  = complete reduction of itch; additionally free text options to indicate specific creams, tablets or alternative medicine)
preferred treatment options | single time point assessment at baseline
  Questions regarding preferred treatment options (NRS 0- 10; 0 = unimportant, 10 = most important; including additional free text option)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Müller, Dr. med, Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (1):
- Department of Dermatology, University Hospital Basel, Basel, Switzerland